CLINICAL TRIAL: NCT01859000
Title: Family-Based Drug Services for Young Disaster Victims
Acronym: Katrina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cynthia Rowe, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 20057675; R01DA021887 (NIH)
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Substance Abuse; Families; Trauma
Keywords: Adolescents; Hurricane Katrina; Family-based treatment; Multidimensional Family Therapy; Group CBT
MeSH Terms: conditions — Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidimensional Family Therapy (Experimental): MDFT is a multi-systems family-based approach (Liddle, 2002a) designed to address the multiple developmental disruptions and symptoms that result from interacting individual, family, peer, and community risk factors (Liddle, 2002a). MDFT assesses and intervenes at multiple levels and in multiple domains of the adolescent's life -- individual, familial and extrafamilial.
  Interventions: Other: Multidimensional Family Therapy
- Group CBT (Other): The group treatment employed in the proposed study is a state-of-the-art peer group-based CBT model. The treatment will be based on established guidelines for CBT therapy for teen substance abuse (CSAT, 1999; Waldron & Kaminer, 2004) as well as trauma (La Greca & Silverman, in press). The treatment adopts a risk and protective factor framework, seeking to reduce substance use both by targeting cognitions about use directly and by focusing on accompanying problem behaviors such as poor academic performance and limited social skills (Hawkins et al, 1992).
  Interventions: Other: Group CBT

INTERVENTIONS:
Other: Multidimensional Family Therapy — MDFT assesses and intervenes in four domains to address comorbid substance abuse and trauma symptoms: 1) adolescent, 2) parent, 3) family, and 4) external systems. MDFT therapists will address trauma symptoms among both teens and parents, aiming to improve coping and reduce the impact of stress on the family. Consistent with a multidimensional approach, MDFT trauma-focused interventions address the needs of both youth and their parents, and MDFT therapists seek collaboration and advocacy from school and court personnel.
  Other Names: MDFT
  Arms: Multidimensional Family Therapy
Other: Group CBT — Trauma symptoms will be addressed using techniques designed to reduce cognitions that maintain anxiety and depressive symptoms and improve coping, such as cognitive restructuring, gradual exposure, and helping teens to understand and accept reminders of the event and ongoing stressors (Pynoos et al, 1998).
  Arms: Group CBT

SUMMARY:
This protocol seizes this rare scientific opportunity to test an integrative family based model to address youths' coexisting substance abuse and trauma in the wake of Hurricane Katrina. The study would address a number of gaps in the current evidence base related to understanding and treating comorbid teen drug abuse and trauma that may be initiated or exacerbated in the wake of disasters such as Hurricane Katrina. This study would compare two promising interventions for youth with comorbid trauma and substance abuse, family-based treatment and group Cognitive Behavioral Therapy (CBT), potentially yielding new and vital information about effective treatment for substance abusing youth following traumatic events.

DETAILED DESCRIPTION:
This study is a 2 (treatments) by 5 (time points), repeated measures intent-to-treat randomized control design with multiple dependent variables. The sample includes a total of 150 ethnically diverse adolescents who are clinically referred for substance abuse treatment throughout St. Charles Parish, a New Orleans area parish that was heavily impacted by Hurricane Katrina. The parish has high rates of teen substance abuse as documented in school surveys (State of Louisiana Office for Addictive Disorders, 2002, 2004). Eligible youth, who meet American Society of Addiction Medicine (ASAM) criteria for outpatient substance abuse treatment and report trauma symptoms related to Hurricane Katrina, will be randomized to a family-based treatment (MDFT) or group CBT. Both treatments will be delivered approximately twice weekly over 4 months. Assessments of youth and family functioning across several domains will be conducted at intake, 2, 4, 6, and 12 month follow-up. Measuring multiple domains at several assessment points within and following treatment (Brown, 2004) will enable investigators to examine trajectories of change as well as mediators and moderators of treatment effects.

The study has four aims:

Aim 1: To explore links between hurricane-related stress and trauma and youths' substance abuse.

Hypothesis 1: Severity of youths' substance use at intake to treatment will be predicted by level of exposure to Hurricane Katrina, stressful life events following Katrina, trauma symptoms, and coping.

Aim 2: To investigate in a community based randomized control trial the effectiveness of a family-based intervention (MDFT) vs. group CBT for teen substance abusers impacted by Hurricane Katrina.

Hypothesis 2a: Family-based treatment (MDFT) will more effectively reduce youths' substance abuse, delinquency, trauma, and school problems up to one year post-intake than a group CBT approach.

Hypothesis 2b: Family-based treatment (MDFT) will more effectively reduce parents' stress and family conflict up to one year post-intake than group CBT.

Hypothesis 2c: Youth assigned to MDFT will be less likely to meet diagnostic criteria for PTSD at 12 month post-intake than group CBT.

Aim 3: To examine teen and parent coping as mediators of treatment effects.

Hypothesis 3a: Youth in MDFT will develop more effective coping strategies than those in group CBT through improved parental coping and parenting practices, and lower family conflict, as well as directly through intervention effects.

Hypothesis 3b: Youth in MDFT will achieve greater reductions in substance abuse and trauma symptoms than those in group treatment through more effective coping during the 12 month follow-up period.

Aim 4: To explore moderators of treatment effects based on post-Katrina stress and trauma symptoms.

Hypothesis 4: The advantage of MDFT over group CBT in decreasing substance abuse will be more pronounced with youth who report higher levels of disaster-related stress and trauma symptoms at intake.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 13 and 17
* Meet ASAM criteria for outpatient substance abuse treatment
* At least mild trauma symptoms on PTSD-Reaction Index
* Not receiving any other behavioral treatment
* Parent/guardian willing to participate in the study/treatment
* Parent informed consent and youth informed assent to participate in the study

Exclusion Criteria:

* Mental retardation or pervasive developmental disorders
* Psychotic disorder as indicated by record review
* current suicidality as indicated by verbalization of ideation + intent + plan in interview

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2007-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Substance use | Intake through the 12-month follow-up
  The Timeline Follow-Back Method, Personal Experiences Inventory and Urinalyses will be used to measure substance use.

SECONDARY OUTCOMES:
Delinquency | One year prior to intake through the 12-month follow-up
  Court records and the National Youth Survey Self-Report Delinquency Scale (SRD)will be used to assess delinquency.
Trauma Symptoms | Screening through the 12-month follow-up
  Posttraumatic Stress Disorder Reaction Index Revised will be used to measure trauma symptoms with youth.
School Problems | One year prior to intake through the 12-month follow-up
  School records will be obtained for each youth enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rowe, Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - The Center for Family and Youth Services, Luling, Louisiana

REFERENCES:
- [Background] Rowe CL, La Greca AM, Alexandersson A. Family and individual factors associated with substance involvement and PTS symptoms among adolescents in greater New Orleans after Hurricane Katrina. J Consult Clin Psychol. 2010 Dec;78(6):806-817. doi: 10.1037/a0020808. PMID 20919759